CLINICAL TRIAL: NCT06237465
Title: Botulinum Toxin-A for Hidradenitis Suppurativa
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never officially began (or enrolled)
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000034975; 000 (Other: CTGTY)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa; Hidradenitis Suppurativa (HS); Hidradenitis Suppurativa, Acne Inversa
Keywords: hidradenitis suppurativa; Botulinum Toxin-A
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Saline Solution; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): During their treatment visit, subjects will receive Botulinum Toxin-A in one axillae and normal saline in the other, in a double-blinded fashion.
  Interventions: Drug: Botulinum toxin type A
- Placebo Comparator (Placebo Comparator): At three months, Group 1 subjects will receive 50-units BTX-A and NS in the same axillae as before while Group 2 will receive NS in both axillae.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Thirty subjects with active bilateral axillary hidradenitis suppurativa will be consecutively enrolled and randomly stratified into two groups (Group 1 and Group 2). Both groups will contain five subjects each with mild, moderate, and severe disease. All participants will have 50-units of Botulinum Toxin-A (BTX-A) injected intradermally in one axilla and normal saline (NS) placebo administered in the other in a randomized, double-blinded fashion. At three months, Group 1 will receive 50-units BTX-A and NS in the same axillae as before while Group 2 will receive NS in both axillae.
  Other Names: Placebo
  Arms: Placebo Comparator
Drug: Botulinum toxin type A — Thirty subjects with active bilateral axillary hidradenitis suppurativa will be consecutively enrolled and randomly stratified into two groups (Group 1 and Group 2). Both groups will contain five subjects each with mild, moderate, and severe disease. All participants will have 50-units of Botulinum Toxin-A (BTX-A) injected intradermally in one axilla and normal saline (NS) placebo administered in the other in a randomized, double-blinded fashion. At three months, Group 1 will receive 50-units BTX-A and NS in the same axillae as before while Group 2 will receive NS in both axillae.
  Arms: Experimental

SUMMARY:
The purpose of this research study is to determine if the medication Botulinum Toxin-A (BTX-A) is effective in treating hidradenitis suppurativa (HS)

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is an auto-inflammatory disorder of apocrine sweat glands which results in painful, draining nodules within hair-bearing skin of the axillae, groin, and perineum. There is no consensus for treatment of HS and neither a medical nor surgical cure exists. Several case reports show potential efficacy of Botulinum Toxin-A (BTX-A) in inducing remission of HS however, these studies are underpowered. The objective of this study is to determine if Botulinum Toxin- A induces regression, remission, or relapse of hidradenitis suppurativa lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active axillary hidradenitis suppurativa of the same severity bilaterally. regimen
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* Agreement to forego other treatments for hidradenitis for the duration of the study

Exclusion Criteria:

* Current use of antibiotics, hormonal therapies, steroids, and/or biologics
* Presence of cardiac pacemaker
* Pregnancy or lactation
* Known neuromuscular disorder
* Known hyperhidrosis
* Febrile illness within one month
* Treatment with another investigational drug or other intervention within three months
* Patients without active axillary hidradenitis suppurativa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Number of lesions | baseline and 3 months
  Change in number of lesions (nodules, abscesses, and fistulous tracts). Any changes in lesion count or size will be documented and subjective symptoms such as pain will be noted.

SECONDARY OUTCOMES:
Change in Hidradenitis Suppurativa Quality of Life (HiSQOL) score | baseline, 3 months and 6 months
  HiSQOL is a patient-reported outcome measure developed for clinical trials to address disease-specific changes in HR quality of life (HRQOL). The item scores are summed to create a total ranging from 0 to 68, with higher scores indicating more severe impact on HRQOL.
Change in Duration of Effect of BTX-A in Hidradenitis Suppurativa | 3 months, 6 months, 12 months
  Subjects will be clinically evaluated at 3, 6, and 12 months to monitor qualitative and quantitative change in lesions (nodules, abscesses, fistulous tracts) and symptoms (pain, drainage, swelling, and impairment) and duration of change, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Rummana Aslam, MD, Principal Investigator — Department: Orthopedics and Rehabilitation, Yale New Haven Hospital, Yale School of Medicine, Yale University
Locations (1):
- Yale Medicine Multispecialty Clinic, Guilford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horowitz LM, Snyder DJ, Boudreaux ED, He JP, Harrington CJ, Cai J, Claassen CA, Salhany JE, Dao T, Chaves JF, Jobes DA, Merikangas KR, Bridge JA, Pao M. Validation of the Ask Suicide-Screening Questions for Adult Medical Inpatients: A Brief Tool for All Ages. Psychosomatics. 2020 Nov-Dec;61(6):713-722. doi: 10.1016/j.psym.2020.04.008. Epub 2020 Apr 28. PMID 32487323
- [Background] Hua VJ, Kuo KY, Cho HG, Sarin KY. Hyperhidrosis affects quality of life in hidradenitis suppurativa: A prospective analysis. J Am Acad Dermatol. 2020 Mar;82(3):753-754. doi: 10.1016/j.jaad.2019.08.046. Epub 2019 Aug 23. No abstract available. PMID 31449904
- [Background] Campanati A, Martina E, Giuliodori K, Bobyr I, Consales V, Offidani A. Two cases of Hidradenitis suppurativa and botulinum toxin type a therapy: A novel approach for a pathology that is still difficult to manage. Dermatol Ther. 2019 May;32(3):e12841. doi: 10.1111/dth.12841. Epub 2019 Feb 10. PMID 30693648
- [Background] Shi W, Schultz S, Strouse A, Gater DR. Successful treatment of stage III hidradenitis suppurativa with botulinum toxin A. BMJ Case Rep. 2019 Jan 20;12(1):e226064. doi: 10.1136/bcr-2018-226064. PMID 30665927
- [Background] Khoo AB, Burova EP. Hidradenitis suppurativa treated with Clostridium botulinum toxin A. Clin Exp Dermatol. 2014 Aug;39(6):749-50. doi: 10.1111/ced.12380. Epub 2014 Jul 1. No abstract available. PMID 24986398
- [Background] Feito-Rodriguez M, Sendagorta-Cudos E, Herranz-Pinto P, de Lucas-Laguna R. Prepubertal hidradenitis suppurativa successfully treated with botulinum toxin A. Dermatol Surg. 2009 Aug;35(8):1300-2. doi: 10.1111/j.1524-4725.2009.01231.x. Epub 2009 Jun 3. No abstract available. PMID 19496796
- [Background] O'Reilly DJ, Pleat JM, Richards AM. Treatment of hidradenitis suppurativa with botulinum toxin A. Plast Reconstr Surg. 2005 Oct;116(5):1575-6. doi: 10.1097/01.prs.0000184354.32111.dc. No abstract available. PMID 16217533
- [Background] Ravi M, Trinidad J. Botulinum Toxin in Hidradenitis Suppurativa: A Systematic Review. J Drugs Dermatol. 2022 Apr 1;21(4):408-412. doi: 10.36849/JDD.5747. PMID 35389587
- [Background] Grimstad O, Kvammen BO, Swartling C. Botulinum Toxin Type B for Hidradenitis Suppurativa: A Randomised, Double-Blind, Placebo-Controlled Pilot Study. Am J Clin Dermatol. 2020 Oct;21(5):741-748. doi: 10.1007/s40257-020-00537-9. PMID 32761500